CLINICAL TRIAL: NCT06328634
Title: Bacillus Cereus : a Retrospective Study of Patients Diagnosed at Nîmes University Hospital With a Positive Culture for B. Cereus From January 1, 2008 and Literature Review
Brief Title: Bacillus Cereus Infection of Patients Diagnosed at Nîmes University Hospital
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/FV-01
Record Dates: First submitted 2017-02-02; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Bacillus Cereus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
OBJECTIVES:

We aimed to study the characteristics of patients presenting with a Bacillus cereus infection in a university hospital.

METHODS:

We performed a retrospective analysis of the clinical, biological, and treatment-related data of patients hospitalized in our university hospital between January 1st, 2008 and December 31st, 2012 and diagnosed with a B. cereus infection. We identified a subgroup of patients presenting with bacteremia and looked for risk factors for death within that group of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with a B. cereus infection
* patients adult (>18)

Exclusion Criteria:

* patientn diagnosed without infection by B. Cereus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with a B. cereus infection who were hospitalized in our university hospital between January 1st, 2008 and December 31st, 2012.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
descriptive analysis of patients' characteristics and B. cereus infection or colonization. | 4 years

REFERENCES:
- [Result] Veysseyre F, Fourcade C, Lavigne JP, Sotto A. Bacillus cereus infection: 57 case patients and a literature review. Med Mal Infect. 2015 Nov-Dec;45(11-12):436-40. doi: 10.1016/j.medmal.2015.09.011. Epub 2015 Oct 31. PMID 26525185